CLINICAL TRIAL: NCT00653770
Title: A Phase I Study to Assess the Safety and Immunogenicity of New TB Vaccine Candidates FP85A and MVA85A, in Healthy Adults Who Have Previously Been Immunized With BCG, Using a Prime-boost Delivery Schedule
Brief Title: A Phase I Study to Assess the Safety and Immunogenicity of Tuberculosis (TB) Vaccine Candidates FP85A and MVA85A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Dr Helen McShane, University of Oxford
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TB017
Record Dates: First submitted 2008-04-02; First posted 2008-04-07 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2010-02

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — MVA 85A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): FP85A at day 0
  Interventions: Biological: FP85A
- 2 (Experimental): MVA85A at day 0 and FP85A at day 28
  Interventions: Biological: FP85A; Biological: MVA85A
- 3 (Experimental): FP85A at day 0 and MVA85A at day 28
  Interventions: Biological: FP85A; Biological: MVA85A

INTERVENTIONS:
Biological: FP85A — Recombinant Fowlpox virus 9 expressing antigen 85A from M. tuberculosis (5 x10^7 pfu)
Biological: MVA85A — Modified vaccinia virus Ankara expressing antigen 85A from M. tuberculosis (5 x 10^7 pfu)
  Arms: 2; 3

SUMMARY:
This is a Phase I study whose primary outcome is to assess the safety of a new tuberculosis vaccine, FP85A, when administered individually and sequentially with MVA85A in a prime-boost regime, to healthy volunteers, who have previously been vaccinated with BCG. The secondary outcome is to assess the cellular immune response in the same population. The trial consists of 36 subjects in 3 groups. The first group will be vaccinated with FP85A alone, the second group will be vaccinated with MVA85A followed by FP85A 28 days later and the third group will be vaccinated with FP85A followed by MVA85A 28 days later.

DETAILED DESCRIPTION:
Recombinant fowlpox virus as a vector

Fowlpox virus is only infectious to avian species, but it is able to express antigens in mammalian cells and induce protective immune responses, making it a suitable candidate vector. Recombinant fowlpox viruses have been developed that express antigens from tumour cells, HIV and malaria. FP9 is a live, highly attenuated form of a European strain of fowlpox virus. It was derived from multiple passages in avian cells, followed by plaque purification and the genome has been fully characterised. Fowlpox virus was initially used as a recombinant avian vaccine, but it has also been shown to be a potent inducer of CD8+T cells in preclinical mammalian models and in human trials . In fact, FP9 was found to be more immunogenic than wild type fowlpox and, when used with recombinant MVA in a prime boost regime induced a protective immune response against Plasmodium berghi.

Clinical experience with recombinant fowlpox viruses in Oxford Three FP vaccines encoding different malaria antigens have been used so far in clinical trials in Oxford, FP9 ME-TRAP, FP9 CS and FP9 PP. To date 87 doses of FP9 ME-TRAP have been given to 55 volunteers in Oxford using various regimens in combination with DNA as well as recombinant MVA vaccines. The local and systemic safety profile of FP9 ME-TRAP is comparable to that described for recombinant MVA vaccines. No vaccine-related serious adverse events have been observed. Pain and erythema at the injection site are the predominant local side effects, with the erythema being maximal within 2 to 3 days post-vaccination before receding. The commonest systemic side effect after FP9 ME-TRAP is of feeling feverish although this is not always associated with a documented fever. Other solicited side effects are myalgia, arthralgia, headache and nausea. FP9 CS has been used recently in a phase I study in 25 healthy volunteers in Oxford, at doses of 1x10^8 pfu. Analysis of safety and tolerability suggests similar side effect profile to FP9 ME-TRAP. No serious adverse events were noted in the study. In a phase I/IIa study which is nearing completion, 15 volunteers were immunised with 5x10^7 pfu of FP9 PP, with no vaccine-related serious adverse events and comparable adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged 18 to 50 years
* Resident in or near Oxford for the duration of the vaccination study
* Immunization with BCG greater than 12 months prior to enrolment in the study
* Able and willing (in the Investigators' opinions) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner
* Agreement to practice barrier contraception from the start of the study until 3 months after the final vaccination
* For females, a negative pregnancy test on the day of vaccination and agreement to practice effective contraception for the entire duration of the study
* Agreement to refrain from blood donation during the course of the study
* Written informed consent

Exclusion Criteria:

* Participation in another research study involving an investigational product in the 30 days preceding enrolment, or planned use during the study period
* Prior receipt of a recombinant MVA or fowlpox vaccine
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g. egg products
* Any history of anaphylaxis in reaction to vaccination
* Close contact with fowl during the study period (e.g. chicken farming)
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of serious psychiatric condition
* Any other chronic illness requiring hospital specialist supervision
* Suspected or known current injecting drug or alcohol abuse (as defined by an alcohol intake of greater than 42 units every week)
* Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for hepatitis C virus (antibodies to HCV)
* For females, pregnancy, lactation or willingness/intention to become pregnant during the study
* Any other significant disease, disorder or finding, which, in the opinion of the Investigators, may either put the volunteer at risk because of participation in the study, or may influence the result of the study, or the volunteer's ability to participate in the study.
* Mantoux skin test equal to or greater than 15 millimetres
* Screening Elispot positive (greater than 17 sfc/million PBMC) in any ESAT6 peptide or CFP10 peptide pool
* Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2007-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To assess the safety of a new tuberculosis vaccine, FP85A, when administered individually and sequentially with MVA85A in a prime-boost regime, to healthy volunteers, who have previously been vaccinated with BCG | 3 months

SECONDARY OUTCOMES:
To assess the cellular immune response generated by FP85A, when administered individually and sequentially with MVA85A in a prime-boost regime to healthy volunteers, who have previously been vaccinated with BCG. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Helen McShane, Principal Investigator — University of Oxford
Locations (1):
- CCVTM, University of Oxford, Oxford, United Kingdom

REFERENCES:
- [Derived] Rowland R, Pathan AA, Satti I, Poulton ID, Matsumiya MM, Whittaker M, Minassian AM, O'Hara GA, Hamill M, Scott JT, Harris SA, Poyntz HC, Bateman C, Meyer J, Williams N, Gilbert SC, Lawrie AM, Hill AV, McShane H. Safety and immunogenicity of an FP9-vectored candidate tuberculosis vaccine (FP85A), alone and with candidate vaccine MVA85A in BCG-vaccinated healthy adults: a phase I clinical trial. Hum Vaccin Immunother. 2013 Jan;9(1):50-62. doi: 10.4161/hv.22464. Epub 2012 Nov 10. PMID 23143773